CLINICAL TRIAL: NCT03106974
Title: A Comparison of Tracheal Intubation Using the Totaltrack vs the Macintosh Laryngoscope
Brief Title: A Comparison of Tracheal Intubation Using the Totaltrack vs the Macintosh Laryngoscope in Obese Patients
Acronym: Ovesion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: AnestesiaR (Other)
Responsible Party: Principal Investigator, Eugenio Martinez Hurtado, Principal Investigator, AnestesiaR
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: totaltrackeca01
Record Dates: First submitted 2017-03-26; First posted 2017-04-11 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Endotracheal Intubation; Obesity; Desaturation; Ventilation
MeSH Terms: conditions — Obesity; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Macintosh Laryngoscope (Active Comparator): orotracheal intubation (OTI) with Macintosh Laryngoscope Direct laryngoscopy
  Interventions: Device: orotracheal intubation Macintosh Laryngoscope
- Totaltrack VLM (Active Comparator): orotracheal intubation (OTI) with Totaltrack VlM Indirect laryngoscopy
  Interventions: Device: orotracheal intubation Totaltrack VLM

INTERVENTIONS:
Device: orotracheal intubation Macintosh Laryngoscope — orotracheal intubation (OTI) after induction of anesthesia and complete relaxation
  Other Names: OTI
  Arms: Macintosh Laryngoscope
Device: orotracheal intubation Totaltrack VLM — orotracheal intubation (OTI) after induction of anesthesia and complete relaxation
  Arms: Totaltrack VLM

SUMMARY:
Airway management in obese patients has to consider that mask ventilation (DMV) risk is increased and difficult tracheal intubation (DTI) risk may be increased too.

In obese patients, is essential to prevent early arterial oxygen desaturation related to a reduced functional residual capacity (FRC), atelectasis formation during anesthetic induction and after tracheal intubation, because oxygenation maintenance is the cornerstone of the airway management of the obese patient.

Endotracheal intubation is usually required to allow unrestricted surgical approach. The Macintosh laryngoscope is the standard method. However, sometimes this technique is ineffective and poorly tolerated by the obese patient.

The Totaltrack™ (MedComflow S.A., Barcelona, Spain) is a hybrid device, between a supraglottic airway and a videolaryngoscope with an anatomically shaped blade. It allows fibreoptic visualization of the larynx for tracheal intubation and was developed to aid both ventilation and tracheal intubation, at the time of anticipated and unanticipated difficult airway management.

However, despite its use in clinical practice, there are no comparative studies regarding direct laryngoscopy in obese patients.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 30.
* ASA 1-3
* Scheduled surgeries that require orotracheal intubation.
* General anesthesia with neuromuscular relaxation before intubation.
* Patients who sign informed consent.

Exclusion Criteria:

* ASA 4
* Difficult airway already known.
* Alterations of airway documented, with previous tracheostomy or involve anatomical alterations.
* General anesthesia that not require orotracheal intubation or neuromuscular relaxation.
* Symptomatic gastro-esophageal reflux.
* Lap-Band carrier.
* Allergy medications to use.
* Urgent surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1440 (Estimated)
Dates: Start 2017-05-01 (Estimated); Primary Completion 2018-05-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
saturation of blood oxygen at the end of orotracheal intubation | Time of Orotracheal intubation (TOTI) (up to 1 hour)
  We will compare the blood oxygen saturation at the end of orotracheal intubation with macintosh and totaltrack.
  The end of successful tracheal intubation will be established to obtain a curve of Capnography.

SECONDARY OUTCOMES:
Total time of successful intubation | Time of Orotracheal intubation (TOTI) (up to 1 hour)
  Total time of successful intubation
number of maneuvers | Time of Orotracheal intubation (TOTI) (up to 1 hour)
  number of maneuvers
IDS Scale | Time of Orotracheal intubation (TOTI) (up to 1 hour)
  IDS Scale
POGO Score | Time of Orotracheal intubation (TOTI) (up to 1 hour)
  POGO Score
Number of attempts of endotracheal intubation | Time of Orotracheal intubation (TOTI) (up to 1 hour)
  Number of attempts of endotracheal intubation
hemodynamic response | TOTI pre and postintubation (up to 10 minutes)
  hemodynamic response
Degree of satisfaction of the researcher | time of postintubation (up to 10 minutes)
  Visual Analogic Scale (0-5)
adverse effects encountered during intubation | Time of Orotracheal intubation (TOTI) (up to 1 hour)
  adverse effects encountered during intubation
Complications | Time Frame: TOTI and postintubation (up to 24 hours)
  Complications after intubation

CONTACTS AND LOCATIONS:
Overall Officials: Maria Luisa Mariscal Flores, M.D., Principal Investigator — Hospital Universitario Getafe; Míriam Sánchez Merchante, M.D., Principal Investigator — Hospital Universitario Fundación Alcorcón; Sergio D. Bergese, M.D., Principal Investigator — Clinical Faculty - Wexner Medical Center at The Ohio State University
Locations (1):
- Hospital Universitario Infanta Leonor, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided